CLINICAL TRIAL: NCT03354936
Title: A Multicenter Observational Cohort for HIV Infected Patients With a Cancer Treated by Immune-Checkpoint Inhibitors.
Brief Title: ANRS CO24 OncoVIHAC (Onco VIH Anti Checkpoint)
Acronym: OncoVIHAC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: Pitié-Salpêtrière Hospital (Other); Bicetre Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-A00699-44
Record Dates: First submitted 2017-09-21; First posted 2017-11-28 (Actual); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: HIV Infected Patients With Cancer Treated by ICPi
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — No intervention in the observatory, a collection of data will be carried out in M0, M6, M12, M18 and M24.
  For the physiopathological Substudy OncoVIRIM : Blood samples will be collected to constitute cell bank, plasma bank, serum bank, DNA bank in order to meet the objectives of this substudy and possibly for complementary research.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: Blood sample — Blood samples will be collected to constitute cell bank, plasma bank, serum bank, DNA bank in order to meet the objectives of this substudy and possibly for complementary research

SUMMARY:
A Multicenter, Observational, National Cohort for HIV Infected Patients with a Cancer treated by Immune-Checkpoint Inhibitors (ICPi) for less than one month or to be treated with an ICPi such as anti-PD-1 or anti-PDL-1 or anti-CTLA4, monitored in some French hospitals .

The objective of the study is to assess the safety of these new agents in HIV-infected patients.

As an observatory, the number of participants planned is not predetermined: the aim is to include for 2 years any participant infected with HIV and having a cancer treated by ICPi in one of the centers that have agreed to participate.

50 participants will be recruited for Substudy "OncoVIRIM" during the study period (regardless of tumor type or ICPi type); 8 or 9 time points (blood samples) will be scheduled

The cohort " ANRS CO24 OncoVIHAC " is declared to authorities like category 2 research .

No intervention in the observatory, a collection of data will be carried out in M0, M6, M12, M18 and M24.

For the physiopathological Substudy OncoVIRIM : Blood samples will be collected to constitute cell bank, plasma bank, serum bank, DNA bank in order to meet the objectives of this substudy and possibly for complementary research

DETAILED DESCRIPTION:
Primary Objective To evaluate clinical and biological safety of the use of immune checkpoint inhibitors in HIV infected patients with cancer treated by Immune-Checkpoint Inhibitors (ICPi).

Secondary objectives

* To evaluate evolution of HIV immunological and virological data in HIV infected patients with cancer treated by Immune-Checkpoint Inhibitors (ICPi):
* HIV-RNA plasma viral load
* Evolution of CD4+ and CD8+ T cells counts, CD4/CD8 ratio
* To assess the efficacy endpoint : progression-free survival, overall survival rate at 1 year and 2 years.
* Potential Modification of antiretroviral therapy

Secondary objectives of the Physiopathological Substudy "OncoVIRIM" (Limited to a few clinical centers with a suitable technical tray) :

* To evaluate response to ICPi treatment according to RECIST criteria (solid tumor) and CHESON criteria (lymphoma)
* Other immunological and virological explorations on HIV :
* To evaluate low level HIV replication and size of the HIV reservoir
* To evaluate effects of ICPi on HIV-specific immune responses
* To show the effects of ICPi on HIV-related immune alterations such as T cell differentiation, T cell activation/exhaustion and systemic inflammation
* To demonstrate an effect on other viruses-specific T cells and viremia (EBV, CMV, HHV-8, HBV et HCV (if co-infected)
* To better understand the pathophysiology of ICPi-related immune adverse effects, particularly the development of infraclinical auto-immunity : monitoring of autoantibodies and analysis of changes in B cell antibodies repertoires
* To find immune biomarkers predictive for clinical response to ICPi, MHC class I and II in particular and description of any gene of interest in the context of ICPi treatment

ELIGIBILITY:
Study Population for Cohort

Inclusion criteria :

* Age ≥ 18 years
* Documented HIV-1 infection treated or untreated with antiretrovirals
* Cancer histologically and /or cytologically proven
* Person treated for less than 30 days or who should be treated with anti-PD-1 or anti-PDL-1 or anti-CTLA4 according to current recommendations
* Signed informed consent

Exclusion Criteria

- Subject participating in clinical trials "CHIVA 2" (Lung Cancer- IFCT) and "HANOVRE" (Hodgkin's disease - LYSA)

Study Population for the Physiopathological Substudy "OncoVIRIM":

Inclusion criteria:

* Participant included in the observatory
* Stable antiretroviral therapy (ART) with controlled HIV-RNA plasma viral load ≤ 50 copies/mL
* Beneficiary of a Social Security program (State Medical Aid or AME is not a Social Security program), article L1121-11 of the Public health code…
* Signed informed consent.

Non Inclusion Criteria

* Brain or lung radiotherapy < 30 days
* Transplant organ or bone marrow transplant
* Corticosteroid > 10 mg per day
* Participant who started ICPi treatment prior to inclusion in the observatory

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV Infected Patients with a Cancer treated by Immune-Checkpoint Inhibitors.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-01-17 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-06-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of clinical and biological adverse events occurring with ICPi treatment during the study period | 4.5 years

SECONDARY OUTCOMES:
Immuno-virological evolution | between Month0 and Month24
  HIV-RNA plasma viral load copies/mL
Immuno-virological evolution | between Month0 and Month 24
  CD4+ and CD8+ T cells counts /mm3 and %, CD4/CD8 ratio.
Disease status | at Month12 and at Month24
  Overall response rate
Progression-Free survival | at Month6, Month12, Month18, Month24
  Progression-Free survival rate
For Physiopathological Substudy "OncoVIRIM" : Objective Response Rate (OPR) | At following cures cycles according to the type of treatment : Cycle1 (Week0), Cycle2 (Week2 or Week3), Cycle3 (Week4 or Week6), Cycle9 (Week16) or Cycle9 (Week24), Cycle 15(Week28), Cycle18 (Week52), Cycle27 (Week52), Cycle36 (Week104), Month6, Month12
  Objective response rate of patient tumor with ICPi treatment according to RECIST criteria (solid tumor) et CHESON criteria (lymphoma).
  The cycles of cures concerned according to the type of treatment :
  * Nivolumab with a cure cycle length of 2 weeks : Cycle1(Week0), Cycle2 (Week2), Cycle3 (Week4), Cycle9 (Week16), Cycle15 (Week28), Cycle27 (Week52), Cycle51 (Week100)
  * Pembrolizumab with a cure cycle length of 3 weeks : Cycle1 (Week0), Cycle2 (Week3), Cycle3 (Week6), Cycle9 (Week24), Cycle18 (Week52), Cycle36 (Week104)
  * Ipilimumab with a cure cycle length of 3 weeks : Cycle1 (Week0), Cycle2(Week3), Cycle3 (Week6), Cycle4 (Week9), Month6, Month12
For Physiopathological Substudy "OncoVIRIM" : Detailed Immunological and Virological Evolution | At following cures cycles according to the type of treatment : Cycle1 (Week0), Cycle2 (Week2 or Week3), Cycle3 (Week4 or Week6), Cycle9 (Week16) or Cycle9 (Week24), Cycle 15(Week28), Cycle18 (Week52), Cycle27 (Week52), Cycle36 (Week104), Month6, Month12
  - Low level of HIV-RNA plasma viral load (ultrasensitive assay), HIV-DNA viral load in PBMCs (peripheral blood mononuclear cells)
  The cycles of cures concerned according to the type of treatment :
  * Nivolumab with a cure cycle length of 2 weeks : Cycle1 (Week0), Cycle2 (Week2), Cycle3 (Week4), Cycle9 (Week16), Cycle 15(Week28), Cycle27 (Week52), Cycle51 (Week100), in case of treatment stopped and in case of immunological adverse event.
  * Pembrolizumab with a cure cycle length of 3 weeks : Cycle1 (Week0), Cycle2 (Week3), Cycle3 (Week6), Cycle9 (Week24), Cycle18 (Week52), Cycle36 (Week104) in case of treatment stopped and in case of immunological adverse event.
  * Ipilimumab with a cure cycle length of 3 weeks : Cycle1 (Week0), Cycle2(Week3), Cycle3 (Week6), Cycle4 (Week9), Month 6, Month 12, in case of treatment stopped and in case of immunological adverse event.
For Physiopathological Substudy "OncoVIRIM" : Detailed Immunological and Virological Evolution | At following cures cycles according to the type of treatment : Cycle1 (Week0), Cycle2 (Week2 or Week3), Cycle3 (Week4 or Week6), Cycle9 (Week16) or Cycle9 (Week24), Cycle 15(Week28), Cycle18 (Week52), Cycle27 (Week52), Cycle36 (Week104), Month6, Month12
  - Anti-HIV Specific Immune Responses T cell (polyfunctionality and expression of immune checkpoints)
  The cycles of cures concerned according to the type of treatment :
  * Nivolumab with a cure cycle length of 2 weeks : Cycle1 (Week0), Cycle2 (Week2), Cycle3 (Week4), Cycle9 (Week16), Cycle 15(Week28), Cycle27 (Week52), Cycle51 (Week100), in case of treatment stopped and in case of immunological adverse event.
  * Pembrolizumab with a cure cycle length of 3 weeks : Cycle1 (Week0), Cycle2 (Week3), Cycle3 (Week6), Cycle9 (Week24), Cycle18 (Week52), Cycle36 (Week104) in case of treatment stopped and in case of immunological adverse event.
  * Ipilimumab with a cure cycle length of 3 weeks : Cycle1 (Week0), Cycle2(Week3), Cycle3 (Week6), Cycle4 (Week9), Month 6, Month 12, in case of treatment stopped and in case of immunological adverse event.
For Physiopathological Substudy "OncoVIRIM" : Detailed Immunological and Virological Evolution | At following cures cycles according to the type of treatment : Cycle1 (Week0), Cycle2 (Week2 or Week3), Cycle3 (Week4 or Week6), Cycle9 (Week16) or Cycle9 (Week24), Cycle 15(Week28), Cycle18 (Week52), Cycle27 (Week52), Cycle36 (Week104), Month6, Month12
  - Systemic inflammation markers and markers of T cell activation, exhaustion, and differentiation
  The cycles of cures concerned according to the type of treatment :
  * Nivolumab with a cure cycle length of 2 weeks : Cycle1 (Week0), Cycle2 (Week2), Cycle3 (Week4), Cycle9 (Week16), Cycle 15(Week28), Cycle27 (Week52), Cycle51 (Week100), in case of treatment stopped and in case of immunological adverse event.
  * Pembrolizumab with a cure cycle length of 3 weeks : Cycle1 (Week0), Cycle2 (Week3), Cycle3 (Week6), Cycle9 (Week24), Cycle18 (Week52), Cycle36 (Week104) in case of treatment stopped and in case of immunological adverse event.
  * Ipilimumab with a cure cycle length of 3 weeks : Cycle1 (Week0), Cycle2(Week3), Cycle3 (Week6), Cycle4 (Week9), Month 6, Month 12, in case of treatment stopped and in case of immunological adverse event.
For Physiopathological Substudy "OncoVIRIM" : | between Month0 and Month24
  Incidence of autoimmune complications and changes in antibodies repertoires of B cell in case of immunological adverse event
For Physiopathological Substudy "OncoVIRIM" : Gene sequencing | Week0
  Gene sequencing whose interest appears to be major in the responses / adverse effects of ICPi, especially MHC class I and II

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Philippe SPANO, MD, PhD, Principal Investigator — GH Pitié-Salpêtrière-Charles Foix; Olivier LAMBOTTE, MD, PhD, Principal Investigator — CHU Bicêtre
Locations (56):
- France (56):
  - Service d'Immunologie - Hôpital Felix Guyon, La Réunion, Saint-Denis
  - Service d'Hématologie Oncologie - Centre Hospitalier du Pays d'Aix, Aix-en-Provence
  - Service de pneumologie - Hôpital Victor Dupouy, Argenteuil
  - Service d'Onco-Hématologie Immunodépression - Hôpital Henri Duffaut, Avignon
  - Service des Maladies Infectieuses et Tropicales - Hôpital Jean Minjoz, Besançon
  - Pôle de Médecine 2 - Centre Hospitalier Andrée Rosemon, Cayenne
  - Service de Médecine interne - Hôpital Antoine Béclère, Clamart
  - Service d'hématologie - Hôpital Gabriel Montpied, Clermont-Ferrand
  - Service des Maladies Infectieuses et Tropicales - Hôpital Gabriel Montpied, Clermont-Ferrand
  - Service d'Immunologie Clinique - Hôpital Henri Mondor, Créteil
  - Service de Médecine interne - Centre Hospitalier Intercommunal, Créteil
  - Service de pneumologie - Centre Hospitalier Intercommunal, Créteil
  - Service Hémopathies Lymphoïdes - Hôpital Henri Mondor, Créteil
  - Service Oncologie Médicale - Centre Hospitalier Intercommunal, Créteil
  - Service de Médecine interne et Maladies infectieuses - Hôpital André Mignot, Le Chesnay
  - Service d'hématologie et oncologie - Hôpital André Mignot, Le Chesnay
  - Service de Médecine interne-Immunologie clinique - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - Service des Maladies Infectieuses et Tropicales - Hôpital de la Croix Rousse, Lyon
  - Ambulatoire-Hôpital de Jour - Institut Paoli Calmettes, Marseille
  - Service d'hématologie-Cisih - Hôpital Sainte Marguerite, Marseille
  - Service de dermatologie - Hôpital St Joseph, Marseille
  - Service de Pneumologie - Hôpital St Joseph, Marseille
  - Chirurgie Urologique et Tranplantation Rénale - Hôpital de la Conception, Marseille
  - Service d'Oncologie médicale - Hôpital de la Timone, Marseille
  - Service dermatologie/vénéréologie - Hôpital de la Timone, Marseille
  - Service d'oncologie multidiscliplinaire - Hôpital Nord, Marseille
  - Service de Médecine Interne - Centre Hospitalier de Martigues, Martigues
  - Service des Maladies Infectieuses et Tropicales - Hôpital Gui de Chauliac, Montpellier
  - Service de Dermatologie - Hôpital l'Archet, Nice
  - Service de médecine interne Cancérologie - Hôpital l'Archet, Nice
  - Service des Maladies Infectieuses et Tropicales - Hôpital l'Archet, Nice
  - Service des Maladies Infectieuses - Hôpital Saint Antoine, Paris
  - Service Infectiologie - Hôpital de l'Hôtel-Dieu, Paris
  - Service d'immuno-pathologie clinique - Hôpital Saint-Louis, Paris
  - Service des Maladies Infectieuses - Hôpital Saint-Louis, Paris
  - Servide de Dermatologie - Hôpital Saint-Louis, Paris
  - Service d'Oncologie Médicale - Hôpital Pitié-Salpêtrière, Paris
  - Service des Maladies Infectieuses et Tropicales - Hôpital Pitié-Salpêtrière, Paris
  - Service Hématologie Clinique - Hôpital Pitié-Salpêtrière, Paris
  - Hôpital Bichat, Paris
  - Service d'Immunologie Clinique - Hôpital européen Georges Pompidou, Paris
  - Service de Cancérologie Médicale - Hôpital européen Georges Pompidou, Paris
  - Service de pneumologie - Hôpital Tenon, Paris
  - Service des Maladies Infectieuses et Tropicales - Hôpital Tenon, Paris
  - Service de pneumologie - Hôpital Yves Le Foll, Saint-Brieuc
  - Service Médecine interne - Maladies Infectieuses - Hôpital Yves Le Foll, Saint-Brieuc
  - Service Oncologie Hématologie - Hôpital Yves Le Foll, Saint-Brieuc
  - Centre Hospitalier Universitaire de Saint Etienne, Saint-Priest-en-Jarez
  - Institut de Cancérologie Lucien Neuwirth, Saint-Priest-en-Jarez
  - Le Trait d'Union - Hôpitaux Universitaires de Strasbourg, Strasbourg
  - Service de Médecine Interne - Hôpital Foch, Suresnes
  - Service de Pneumologie - Hôpital Foch, Suresnes
  - Service de Médecine Interne - Hôpital d'Instruction des Armées Saint Anne, Toulon
  - Service des Maladies Infectieuses et Tropicales - Hôpital Purpan, Toulouse
  - Service des Maladies Infectieuses et du Voyageur - Centre Hospitalier de Tourcoing, Tourcoing
  - Département d'Innovation Thérapeutique et d'Essais Précoces - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No